CLINICAL TRIAL: NCT07290413
Title: A Phase 2 Randomized Trial of Intraoral, Extraoral, and Combined Intraoral/Extraoral Photobiomodulation for the Prevention of Oral Mucositis in Patients Undergoing Myeloablative Allogeneic Hematopoietic Cell Transplantation
Brief Title: Photobiomodulation for the Prevention of Oral Mucositis
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Nathaniel Simon Treister, Associate Surgeon, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 25-137
Record Dates: First submitted 2025-12-16; First posted 2025-12-18 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Oral Mucositis
MeSH Terms: conditions — Stomatitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (3):
- Intraoral photobiomodulation (Experimental): Intraoral PBMT device: The THOR intraoral PBMT device emits LED light with an irradiance of 50 mW/cm2 and, when applied for 60 seconds, delivers 3 J/cm2. It is a handheld device with an array of LEDs covered by smooth glass. The therapeutic area is small enough (similar to a popsicle) to place in the mouth comfortably.
  Interventions: Device: Photobiomodulation - INTRAORAL
- Extraoral photobiomodulation (Experimental): Extraoral PBMT device: The extraoral PBMT device is a dual headed probe designed to be connected to the LX2.3 Laser and LED Therapy System. It consists of two high-powered probes designed to emit 850nm light at an intensity of 240 m/cm2. The device is dual-headed in order to treat both sides of the head simultaneously without the need for a sperate control unit.
  Interventions: Device: Photobiomodulation - EXTRAORAL
- Combined intraoral and extraoral photobiomodulation (Experimental): Participants in this arm will receive both intraoral and extraoral photobiomodulation.
  Interventions: Device: Photobiomodulation - INTRAORAL and EXTRAORAL

INTERVENTIONS:
Device: Photobiomodulation - INTRAORAL — Participants will receive intraoral photobiomodulation
  Arms: Intraoral photobiomodulation
Device: Photobiomodulation - EXTRAORAL — Participants will receive extraoral photobiomodulation
  Arms: Extraoral photobiomodulation
Device: Photobiomodulation - INTRAORAL and EXTRAORAL — Participants will receive intraoral and extraoral photobiomodulation
  Arms: Combined intraoral and extraoral photobiomodulation

SUMMARY:
The goal of this clinical trial is to learn if photobiomodulation works to prevent severe oral mucositis in patients who are undergoing allogeneic hematopoietic cell transplantation. The main questions it aims to answer are:

Does 1) intraoral , 2) extraoral, or 3) combined intraoral/extraoral photobiomodulation have optimal prevention/therapeutic effect in prevention of oral mucositis in patients undergoing myeloablative allogeneic hematopoietic stem cell transplantation (alloHSCT).

Participants will:

Be randomized to one of the three treatment arms Receive daily photobiomodulation therapy (from beginning of transplant conditioning through Day +20 after transplantation) Be evaluated for oral mucositis and symptoms daily Visit the clinic once every 2 weeks for checkups and tests Keep a diary of their symptoms and the number of times they use a rescue inhaler

DETAILED DESCRIPTION:
Patients who are planned for alloHSCT will be randomized 1:1:1 to one of the 3 treatment arms, stratified by age (<18, ≥ 18years). This is a phase 2 randomized trial to identify which of the three photobiomodulation therapy (PBMT) devices, 1) intraoral , 2) extraoral, and 3) combined intraoral/extraoral, has optimal prevention/therapeutic effect in prevention of oral mucositis in patients undergoing myeloablative allogeneic hematopoietic stem cell transplantation (alloHSCT). The study will be conducted in parallel, in a quasi-multi-center manner at three other alloHSCT centers (AC Camargo, SP, Brazil; Hospital de Clínicas de Porto Alegre, Porto Alegre, Brazil; Cincinnati Children's Hospital Medical Center; in addition to DFCI/BWH).

Participants will be evaluated daily according to the validated WHO Oral Toxicity Scale by trained and calibrated investigators. Within each arm, a Simon's 2 stage design will be applied in an intention to treat analysis of the proportion of patients who have <5 days of WHO grade ≥ 3 OM, to eliminate arms with insufficient evidence of efficacy. The remaining arms will be analyzed in a selection design (pick the winner) to determine the probability that the arm selected for a future phase 3 trial is either superior to, or at worst, more or less equivalent to, other arm(s). The study will enroll up to 96 patients with up to 26 patients per treatment arm. The accrual rate at DFCI is anticipated to be 2 patients/month, or 24 patients per year. The same accrual rate is anticipated at each of the other three study sites. Therefore, the total accrual of 78 patients can be achieved within 1 year.

The primary endpoint, duration of severe OM, is defined in section 11.1 as the total number of days between day 0 and day +20 on which severe (WHO grade 3 or 4) OM was reported. A conservative approach to missing data will be taken: Any day on which the grading of mucositis is missing will be counted as a day with WHO grade ≥3 OM. Each patient will be classified as either a success or a failure. "Success" will be defined as a patient who has a duration of WHO grade ≥3 OM <5 days; a patient with ≥5 days will be classified as a "failure" (i.e., a binary endpoint).

The secondary endpoints that will be subjectively considered in making the final selection of the winning arm are:

* Adverse events attributed to PBMT administration;
* Patient acceptability of the PBMT administration;
* Operator acceptability of the PBMT administration;
* Duration of time to complete PBMT administration;
* Duration of hospital stay; and,
* Need to initiate parenteral nutrition.

ELIGIBILITY:
Inclusion Criteria:

* Planned to undergo myeloablative allogeneic HCT (with one of the following regimens): FluBu4, FluMel, or CyTBI conditioning and Tac-Mtx GVHD prophylaxis
* Age ≥4 years
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Participants who have had treatment with oral PBMT within four weeks of admission for HSCT.
* Participants who have a history of radiation therapy to the head and neck.
* Participants who have a history of photosensitivity or underlying disease with known photosensitivity.
* Participants who are planned to receive palifermin (keratinocyte growth factor) for OM prevention.
* Participants who have facial hair and unwilling to shave.

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Duration of severe oral mucositis according to the World Health Organization Oral Toxicity Score | Oral mucositis is assessed daily from day 0 through day +20
  WHO Score (0-4, "severe" defined as grades 3 and 4)

CONTACTS AND LOCATIONS:
Locations (1):
- Dana-Farber Cancer Institute, Boston, Massachusetts, United States